CLINICAL TRIAL: NCT01852409
Title: Phase I Trial of Intraperitoneal Bevacizumab in Refractory Malignant Ascites.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGOG6001
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Refractory Malignant Ascites
Keywords: refractory malignant ascites; Bevacizumab; intraperitoneal; phase I
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bevacizumab (Experimental): The study evaluate 4 dose level of bevacizumab:2.5mg /kg;5 mg /kg;7.5mg /kg; 1.25mg /kg;
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab
  Other Names: Avastin

SUMMARY:
Malignant ascites often has a profound impact on the quality of life of cancer patients. Current treatments,including dietary, medical, and procedural are often temporary and unsatisfactory options in patients approaching the end of life. Intraperitoneal bevacizumab for the palliation of malignant ascites might be a novel choice for refractory malignant ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Histologically or cytologically confirmed non-squamous cell carcinoma，including colorectal cancer, gastric cancer, esophageal cancer, pancreatic cancer, bile duct cancer, ovarian cancer, peritoneal primary tumor;Ascites were diagnosed by ultrasound or CT and confirmed malignant ascites by cytology;
3. failed to standard systemic therapy and / or no appropriate treatment for the treatment for malignant ascites
4. Age 18-70 years;
5. Performance Status- Eastern Cooperative Oncology Group (ECOG)≤2;
6. Life expectancy of at least 8 weeks;

Exclusion Criteria:

1. systematic anti-cancer therapy, including chemotherapy (intraperitoneal chemotherapy), radiation therapy, immunotherapy, biological or hormone therapy performed within 2 weeks;
2. tyrosine kinase inhibitors or monoclonal antibodies of anti-vascular endothelial growth factor (VEGF) performed within 4 weeks;
3. Laboratory tests:Absolute neutrophil count<1.0x109/L,Platelet count<75x 109/L,Hemoglobin<8g/dl,PT-INR≥1.5 times upper limit of normal (ULN);Bilirubin≥2 x ULN,AST and ALT≥2.5 times ULN(no liver metastasis),≥5 times ULN(with liver metastasis)Creatinine≥1.5 times ULN or calculated creatinine clearance, using the Cockcroft-Gault formula,<40 mL/min;
4. uncontrolled hypertension:systolic pressure ≥160 mmHg,or diastolic pressure≥100mmHg
5. Known history of severe heart disease,uncontrolled or symptomatic angina, congestive heart failure,clinically significant arrhythmias,myocardial infarction within six months;
6. active (severe or uncontrolled) bleeding (hemorrhage within 3 months> 30 ml), hemoptysis (fresh blood, 4 weeks> 5 ml), bloody ascites
7. thrombosis, tumor thrombus events (including arterial/venous thrombosis, tumor thrombosis, pulmonary embolism, transient ischemic attack)within 12 months;
8. Portal hypertensive disease or severe liver disease, including various types of cirrhosis, obstructive jaundice;
9. concurrent gastrointestinal obstruction, peptic ulcer, Crohn's disease, ulcerative colitis and other gastrointestinal diseases according to investigators' determination that may cause gastrointestinal bleeding or perforation;
10. concurrent severe respiratory disease, or chronic therapy with oxygen or corticosteroids, such as chronic obstructive pulmonary disease, interstitial lung disease, etc.
11. Unresolved or unstable, serious toxicity from prior cancer treatment (any toxicities greater than grade 2 or not recovered from surgery;
12. Symptomatic brain metastasis;
13. Uncontrolled systemic disease,such as infection,unstable diabetes mellitus,etc;
14. Active infection of HIV、HBV、HCV；
15. Major surgery within 4 weeks of start of study treatment, without complete recovery.
16. Pregnant or lactating women.Negative serum pregnancy test (For women of childbearing potential);Fertile patients must use effective contraception.
17. Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF;
18. Received any investigational drug treatment within 4 weeks of start of study treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
adverse events | during the treatment in the hospital,an expected average of 1 week
  participants will be followed for the duration of hospital stay, an expected average of 1 week
Maximum tolerated dose | 1 week
  during the treatment in the hosptital

SECONDARY OUTCOMES:
Objective response rate | 1 week
  ultrasound will be performed every week for efficacy evaluation
time to treatment failure(TTF) | 1 month
  the follow-up visit of time to TTF will be performed every 4 weeks
time to death(TTD) | 2 months
  TTD means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 2 months till death or lost

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Kou F, Gong J, Li Y, Li J, Zhang X, Li J, Shen L. Phase I study of intraperitoneal bevacizumab for treating refractory malignant ascites. J Int Med Res. 2021 Feb;49(2):300060520986664. doi: 10.1177/0300060520986664. PMID 33616416